CLINICAL TRIAL: NCT07281027
Title: Comparing the Effects of Anakinra and Tocilizumab on Outcomes in Patients With New-Onset Refractory Status Epilepticus
Brief Title: COMparison Between Anakinra and Tocilizumab in NORSE - "COMBAT-NORSE"
Acronym: COMBAT-NORSE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Lawrence Hirsch, Professor of Neurology, Yale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000041289; RD-2024C2-39648 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2025-11-21; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: New Onset Refractory Status Epilepticus; New-Onset Refractory Status Epilepticus; Febrile Infection-Related Epilepsy Syndrome (FIRES)
Keywords: refractory status epilepticus; NORSE; FIRES; anakinra; tocilizumab
MeSH Terms: conditions — Status Epilepticus | interventions — Interleukin 1 Receptor Antagonist Protein; tocilizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Randomized Controlled Trial (RCT) Cohort (Active Comparator): A randomized controlled cohort (RCT) of anakinra vs. tocilizumab (targeted immunotherapies) started up to and including 7 days after the onset of status epilepticus (SE)
  Interventions: Drug: Anakinra; Drug: Tocilizumab
- Observational Cohort (Other): An observational cohort enrolling patients with acute cryptogenic NORSE who cannot be randomized or who are identified too late to be randomized by the end of day 7 .
  Interventions: Other: Standard medical treatment

INTERVENTIONS:
Drug: Anakinra — SOC will be followed , Suggested Dose:
  10 mg/kg/day IV, divided into 4 daily doses (q6h) Maximum dose: 400 mg/day
  Arms: Randomized Controlled Trial (RCT) Cohort
Drug: Tocilizumab — SOC will be followed,
  Suggested Dose:
  If <30 kg: 12 mg/kg IV once every 2 weeks If ≥30 kg: 8 mg/kg IV once every 2 weeks Maximum dose: 800 mg per dose
  Arms: Randomized Controlled Trial (RCT) Cohort
Other: Standard medical treatment — For patients who could not be randomized by day 7, standard clinical care will be followed and patients will be followed prospectively and observationally.
  Arms: Observational Cohort

SUMMARY:
The goal of this clinical trial is to find out whether two existing medications-anakinra and tocilizumab-can effectively treat a rare and life-threatening brain condition called NORSE (New-Onset Refractory Status Epilepticus). NORSE causes continuous seizures in previously healthy children and adults and does not respond to standard treatments. It often leads to long-term disability or death.

Doctors currently use anakinra and tocilizumab as second-line treatments when first-line therapies fail, but there is no clear evidence showing which drug works better or when it should be given. This study aims to answer those questions.

The study will enroll patients across 33 hospitals in the United States, Canada, Europe, and Asia.

It includes two groups:

1. Randomized Cohort Patients will be randomly assigned to receive either anakinra or tocilizumab within the first 7 days of their illness. Only patients whose doctors were already planning to use one of these medications as part of standard care will be eligible for randomization. Researchers will monitor their recovery and compare outcomes between the two treatments.
2. Observational Cohort Patients who cannot be randomized-usually because they were diagnosed too late-will still be followed to study how the timing of treatment affects recovery.

Participants will:

* Receive one of the two medications (depending on their group assignment).
* Take part in follow-up assessments over the course of one year, including medical evaluations and surveys. Some participants may be followed annually beyond one year.
* Optionally participate in a 60-minute interview to share their or their caregiver's experience with NORSE.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 and older.
* In their usual state of health prior to their onset of SE.
* Presenting with NORSE as defined in the consensus criteria:

  1. Refractory SE (failed 2 appropriately used anti-seizure medications) in a patient without active epilepsy or other pre-existing relevant neurological disorder and without an acute or active structural, toxic, or metabolic cause found in the first 72 hours.
  2. Includes patients with any RSE, not just super-refractory SE.
  3. Includes patients who ultimately are discovered to have a known etiology (infectious, autoimmune, genetic, etc.), as well as those who remain cryptogenic.

     * Additional Inclusion Criteria for the Randomized Arm:
* Anakinra and/or tocilizumab are being planned or considered as part of standard clinical care.
* The onset of SE was in the prior 7 days at the time of enrollment.

Exclusion Criteria:

* Any acute or active systemic medical illness such as metastatic cancer, renal failure, hepatic failure, poorly controlled diabetes, etc., in the opinion of the investigators. If this is unclear, the study PI Dr. Hirsch will determine if this criterion is met.

Additional Exclusion Criteria for the Randomized Control Cohort:

* Contraindication to either anakinra or tocilizumab as listed in the prescribing information:

  1. Known hypersensitivity to E. Coli-derived proteins, anakinra, tocilizumab, or any component of the products
  2. Active serious infection at the time of initiation
  3. Concomitant use of TNF blocking agents; absolute neutrophil count < 2000; platelet count < 100,000 per mm³; or ALT or AST > 1.5 X the upper limit of normal
  4. Elevated risk of GI perforation.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 438 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale - Extended (GOS-E) | 12 months
  The Glasgow Outcome Scale - Extended (GOS-E) is an 8-point scale used to measure global functional outcome. Participants are scored into one of the 8 categories: 1. Death, 2. Vegetative State, 3. Lower Severe Disability, 4. Upper Severe Disability, 5. Lower Moderate Disability, 6. Upper Moderate Disability, 7. Lower Good Recovery, 8. Upper Good Recovery.

SECONDARY OUTCOMES:
Time to resolution of status epilepticus (SE) | 24 hours off anesthetic drips
  Time (days) until discontinuation of anesthetic drips for 24h for the treatment of SE with no return of SE on EEG
Hospital length of stay | 12 months
  Mean number of days during hospitalization from admission to discharge
Mortality | up to 12 months
  Mortality, number of participants
Number of serious adverse events attributed to anakinra or tocilizumab | From hospitalization to 1 month after stopping treatment, up to 12 months
  Number of serious adverse events attributed to anakinra or tocilizumab
Number of participants Post-NORSE epilepsy | 12 months
  Number of participants with any unprovoked seizures after hospital discharge
Number of participants with Treatment success | 12 months
  Combined measure of lack of need for another immunomodulator after the study drug was begun, plus good outcome at 1 year (GOS-E of 5-8) (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Hirsch, MD, Principal Investigator — Yale University
Locations (33):
- United States (25):
  - Barrow Institute, Phoenix, Arizona
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Children's National (DC), Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Chicago, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - Mass General (MGH), Boston, Massachusetts
  - Beth Israel Deaconess, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska, Lincoln, Nebraska
  - New York University, New York, New York
  - Columbia University, New York, New York
  - Mount Sinai (NY), New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital Philadelphia (CHOP), Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor/Texas Children's, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Western University, London
  - Hospital for Sick Children, Toronto
- Salpêtrière, Paris, France
- University of Modena, Modena, Italy
- Seoul National University Hospital, Seoul, South Korea
- Karolinska Institute, Stockholm, Sweden
- United Kingdom (2):
  - Great Ormond Street Hospital, London
  - King's College, London

IPD SHARING:
Plan to Share IPD: Yes
Making the Full Data Package available to enable other researchers (including PCORI) to use it to re-analyze the data or for independent (i.e., novel) research analyses.